CLINICAL TRIAL: NCT04294030
Title: NOWDx Test for the Diagnosis of Herpes Simplex Virus Type 2
Status: Withdrawn | Type: Observational
Why Stopped: Deprioritized by Sponsor
Sponsor: NOWDiagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NOWDx HSV-2 Study
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: HSV-2 Infection; Herpes Simplex Virus Infection
Keywords: HSV-2; Genital Herpes
MeSH Terms: conditions — Herpes Simplex; Herpes Genitalis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Sexually active persons who self-select for HSV-2 testing: Participants must be a mixture of English and Spanish speaking, geographically diverse, gender diverse, ethnically and racially diverse, economically diverse, and with different levels of education; 18-64 years
  Interventions: Device: Diagnostic Test: NOWDx HSV-2 Test
- Expectant mothers: Participants must be a mixture of English and Spanish speaking, geographically diverse, gender diverse, ethnically and racially diverse, economically diverse, and with different levels of education; 18-64 years
  Interventions: Device: Diagnostic Test: NOWDx HSV-2 Test
- Low prevalence population: Participants must be a mixture of English and Spanish speaking, geographically diverse, gender diverse, ethnically and racially diverse, economically diverse, and with different levels of education; 18-64 years
  Interventions: Device: Diagnostic Test: NOWDx HSV-2 Test
- Lay users: Participants must be a mixture of English and Spanish speaking, geographically diverse, gender diverse, ethnically and racially diverse, economically diverse, and with different levels of education; 18-64 years; 1/2 high risk sexual behavior; 1/2 low risk sexual behavior
  Interventions: Device: Diagnostic Test: NOWDx HSV-2 Test

INTERVENTIONS:
Device: Diagnostic Test: NOWDx HSV-2 Test — For this observational trial, the intervention of interest is the NOWDx HSV-2 Test.

SUMMARY:
This study is designed to compare the performance of the NOWDx HSV-2 Test to a currently marketed device. The intent is to show the rapid test device is comparable to the currently marketed device. The NOWDx HSV-2 Test is intended for qualitatively detecting the presence or absence of human Immunoglobulin G (IgG) class antibodies to HSV-2 in human whole blood to aid in the diagnosis of infection caused by herpes simplex virus type 2 (HSV-2).

DETAILED DESCRIPTION:
The objective of this study is to establish the performance characteristics of the NOWDx HSV-2 Test based on comparison to the HerpeSelect 1 and 2 Immunoblot IgG and HerpeSelect 2 ELISA IgG assays.

The external clinical study along with in-house analytical studies will demonstrate the efficacy of the NOWDx HSV-2 Test as an aid in the diagnosis of HSV-2 infection for at home testing and point of care testing sites. Participants will self test and be tested by Clinical Laboratory Improvement Amendments (CLIA) Waived operators with the NOWDx HSV-2 Test at independent sites in Florida, Kentucky, and Arizona.

Two sample types will be tested with the NOWDx HSV-2 Test for each participant: capillary whole blood and venous whole blood. Sera from each participant will be tested at an independent reference laboratory.

The NOWDx HSV-2 Test will be evaluated in diverse populations of sexually active persons who self-select for genital herpes testing, expectant mothers, and persons claiming to lack sexual experience.

ELIGIBILITY:
* Sexually active persons who self-select for syphilis testing n=750 participants; ~250 per study site Inclusion criteria: sexually active persons 18-64 years old Exclusion criteria: persons <18 years old; persons >64 years old; persons with limited or no reading skills; persons who previously participated in a NOWDx study
* Expectant mothers n=90 participants; ~30 per study site Inclusion criteria: expectant mothers ≥18 years old Exclusion criteria: persons <18 years old; persons with limited or no reading skills; persons who previously participated in a NOWDx study
* Low prevalence population n=201 participants; ~67 per study site Inclusion criteria: persons aged 18-64 years old claiming to lack sexual experience Exclusion criteria: persons <18 years old; persons >64 years old; persons with limited or no reading skills; persons who previously participated in a NOWDx study
* Lay users n=48 participants; ~16 per study site Inclusion criteria: persons 18-64 years old; ½ high risk sexual behavior; ½ low risk sexual behavior Exclusion criteria: persons <18 years old; persons >64 years old; persons with limited or no reading skills; persons who previously participated in a NOWDx study

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Residents of the U.S. who elect to participate in the study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Compare NOWDx HSV-2 Test result to comparator method lab result to assess sensitivity and specificity of investigational device. | through study completion, an average of 6 months
  The results should be presented as sensitivity and specificity as compared to the comparator method and should have a point estimate of 95% with a lower bound of the two-sided 95% confidence interval of 90%.

SECONDARY OUTCOMES:
Compare results of NOWDx HSV-2 Tests conducted by lay users with expected results to evaluate test reproducibility by lay users. | through study completion, an average of 6 months
  Test lay user reproducibility using prepared samples for % agreement with expected results.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Cobb, Principal Investigator — NOW Diagnostics, Inc.
Locations (3):
- United States (3):
  - Clinical Research Consortium, Tempe, Arizona
  - Clinical Research of South Florida, Coral Gables, Florida
  - Alliance for Multispecialty Research Lexington, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No